CLINICAL TRIAL: NCT03636841
Title: Reduction of Operating Time by a Smoke Electroprecipitation Device: Randomized Controlled Study on Laparoscopic Cholecystectomy for Acute Cholecystitis
Brief Title: Reduction of Operating Time by a Smoke Electroprecipitation Device for Acute Cholecystitis
Acronym: Ultravision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-58
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): A group of 30 patients using the new medical device with CE marking (Ultravision ©) switch on
  Interventions: Device: medical device with CE marking (Ultravision ©)
- CONTROL GROUP (Active Comparator): A group of 30 patients using the new medical device with CE marking (Ultravision ©) switch off
  Interventions: Device: medical device with CE marking (Ultravision ©)

INTERVENTIONS:
Device: medical device with CE marking (Ultravision ©) — Ultravision © is a medical device that is used during laparoscopy to reduce the discomfort caused by surgical smoke produced by the electrical section of tissue. It works by using the principle of electrostatic precipitation, that is to say it causes the precipitation of suspended smoke droplets on the organs and walls of the abdomen.

SUMMARY:
The smoke produced by the electric section of the tissues during laparoscopy alters the vision of the operative field and presents potential risks. A new medical device with CE marking (Ultravision ©) has been developed to limit electroprecipitation on the wall and tissues of the abdomen.

The aim of the work is to evaluate the effectiveness of this medical device in laparoscopic cholecystectomy for cholecystitis. It is an intervention for a common pathology where smoke is particularly important due to the tissue inflammation and due to the extensive dissection necessary to perform the surgical procedure.

A randomized double-blinded study will be conducted in two academic hospitals (Marseille North Hospital and Timone, APHM) evaluating the use of a smoke electroprecipitation device (Ultravision ©) during laparoscopic cholecystectomy for cholecystitis operated at the acute phase. A group of 30 patients using the device will be compared to a control group of 30 patients. The evaluation will last thirty days per patient and the duration of inclusion is 2 years.

The main objective is to demonstrate a significant reduction in operating duration by using the device. The secondary objectives are to reduce the CO2 consumption, the surgical incidents and the discomfort of the surgeon related to the smoke.

DETAILED DESCRIPTION:
Context and purpose of the work:

The smoke produced by the electric section of the tissues during laparoscopy alters the vision of the operative field and presents potential risks. A new medical device with CE marking (Ultravision ©) has been developed to limit electroprecipitation on the wall and tissues of the abdomen.

The aim of the work is to evaluate the effectiveness of this medical device in laparoscopic cholecystectomy for cholecystitis. It is an intervention for a common pathology where smoke is particularly important due to the tissue inflammation and due to the extensive dissection necessary to perform the surgical procedure.

Material and method A randomized double-blinded study will be conducted in two academic hospitals (Marseille North Hospital and Timone, APHM) evaluating the use of a smoke electroprecipitation device (Ultravision ©) during laparoscopic cholecystectomy for cholecystitis operated at the acute phase. A group of 30 patients using the device will be compared to a control group of 30 patients. The evaluation will last thirty days per patient and the duration of inclusion is 2 years.

Expected results The main objective is to demonstrate a significant reduction in operating duration by using the device. The secondary objectives are to reduce the CO2 consumption, the surgical incidents and the discomfort of the surgeon related to the smoke.

ELIGIBILITY:
Inclusion Criteria:

* Adult> 18 years old
* Ability to accept consent
* Acute documented cholecystitis (pain> 6h, thickening of vesicular wall on ultrasound, biological inflammatory syndrome)
* Patient operated within 5 days of onset of signs
* Surgery decided by laparoscopy

Exclusion Criteria:

Pregnant woman

* Atcd umbilical abdominal surgery
* Achievement of the open subcostal intervention
* Patient under anticoagulant
* Patient ASA3
* Age <75 years
* BMI> 45
* icteric cholestasis on preoperative laboratory examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
operating time | 2 hours
  the time of the surgery calculated from the incision to the dressing (as is done routinely for each procedure on anesthesia protocols).

CONTACTS AND LOCATIONS:
Overall Officials: emilie garrido pradalie, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France